CLINICAL TRIAL: NCT06689085
Title: Open-Label, Multiple-Dose, 52-Week Study to Evaluate the Safety, PK, & Efficacy of XYOSTED® for Testosterone Replacement in Male Adolescents With Deficiency or Absence of Endogenous Testosterone Due to Primary or Secondary Hypogonadism
Brief Title: 52 Week Study of Safety, PK, & Efficacy of XYOSTED® for Testosterone Replacement in Male Adolescents With Hypogonadism
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATRS QST-19-007
Record Dates: First submitted 2024-11-06; First posted 2024-11-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-05

CONDITIONS: Hypogonadism, Male
Keywords: primary hypogonadism; secondary hypogonadism
MeSH Terms: conditions — Eunuchism; Hypogonadism | interventions — testosterone enanthate; Testosterone Propionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Participants (Experimental): XYOSTED Injection (Testosterone enanthate) 50mg / 0.5 mL, 75 mg/0.5 mL, 100 mg/0.5 mL
  Interventions: Combination Product: Testosterone enanthate

INTERVENTIONS:
Combination Product: Testosterone enanthate — XYOSTED 50mg, XYOSTED 75 mg, XYOSTED 100 mg
  Other Names: XYOSTED Injection

SUMMARY:
This is a 52-week open label single arm study to investigate the effects of XYOSTED, as testosterone replacement therapy, on adolescent males with either primary or secondary hypogonadism.

The study aims to determine the effectiveness of XYOSTED measured by continuation or induction of puberty in addition to XYOSTED dosage, safety and testosterone levels.

DETAILED DESCRIPTION:
This is a Phase 3/4, open-label, multicenter study in approximately 100 males 12 to < 18 years of age with primary or secondary hypogonadism (congenital or acquired). Each participant will be screened for eligibility within 28 days before receiving his first dose of study drug on Day 1. During the Screening period, each participant will have a full clinical examination with pubertal staging (ie, Tanner Stage, Table 11), including 2 separate serum total testosterone (TT) measurements obtained in the early morning, where the average (Cavg) will be considered baseline value. Each participant will be categorized as having primary or secondary hypogonadism prior to dosing on Day 1.

Participants meeting all eligibility criteria will be assigned to a starting dose of XYOSTED based on their weight and Targeted Tanner Stage on Day 1. The Targeted Tanner Stage will be determined during Screening by an experienced pediatric endocrinologist.

Participants will have dose adjustments during the study to achieve their Targeted Tanner Stage. Dose adjustments will be based on reviewing the TT concentration between doses (Cmid) by measuring serum TT 14 days after the administration of XYOSTED for participants receiving the Q4W schedule, and 7 days after the administration of XYOSTED for participants who switch to the Q2W schedule. Participants will be evaluated for further dose adjustments approximately every 3 months to achieve the desired targeted TT level

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with a deficiency or absence of endogenous testosterone due to primary or secondary hypogonadism of a known etiology. Children with combined hormone deficiencies are permitted to enroll (but the child must already be receiving treatment for concomitant hormonal deficiencies)
2. Participants receiving prior testosterone treatment must be receiving a stable dose for at least 12 weeks prior to Screening
3. Have parent(s) or a legal guardian who will voluntarily provide written informed consent for the child to participate in the study
4. Willing to provide assent for participation in the study
5. Be a male 12 to < 18 years of age at the time of consent/assent
6. Have Legally Authorized Representative who is able to understand and comply with all study procedures and agrees to have the child participate in the study program as outlined in the protocol
7. Requires chronic pharmacologic support for the initiation and/or continuation of pubertal maturation
8. Have a body mass index (BMI)-for-age greater than the 5th percentile and weigh ≥ 40 kg
9. If sexually active with a female partner of child-bearing potential, agrees to:

   1. Practice true abstinence including 30 days after the last IP administration, or,
   2. Use 2 adequate forms of highly effective contraception, one of which should be a physical barrier, during the study and for 30 days after the last IP administration.

Exclusion Criteria:

1. Has abnormal thyroid function tests at Screening
2. Has suspected or known constitutional growth delay in growth and puberty (CDGP)
3. Has evidence of possible nutritional or gastrointestinal disorder that may impact growth (e.g., abrupt weight loss within the 3 months prior to Screening, unmanaged celiac disease, inflammatory bowel disease)
4. Has a known allergy or hypersensitivity to XYOSTED, or to any of its ingredients (testosterone enanthate and sesame oil)
5. Participants receiving prior treatment with testosterone who are not on a stable dose for at least 12 weeks prior to Screening.
6. Is receiving testosterone through a transdermal patch or gel in the 12 weeks prior to Screening.
7. Has an allergy to foods or products containing sesame seeds or sesame oil
8. Has Stage 1 hypertension, defined as the average of 2 or more seated right arm BP measurements exceeding the 95th percentile for age, sex, and height, or SBP ≥ 130 mm Hg and/or DBP ≥ 80 mm Hg (Flynn et al., 2017, in Appendix B), at Screening or Day 1.
9. Has a clinically significant abnormal clinical laboratory test value at Screening, as determined by the Investigator including hematocrit ≥ 48%
10. Has a history of deep venous thrombosis or pulmonary embolism
11. Has evidence of a clinically significant 12-lead electrocardiogram (ECG) abnormality at Screening, as determined by the Investigator
12. Has a current suspected or diagnosed (and unresected) tumor of the pituitary gland with the exception of Rathke's cleft cyst or a stable non-functioning pituitary microadenoma (ie, lesion size < 10 mm that has not increased in size over a period of 1 year on repeat imaging), as determined by the Investigator
13. Has an active malignancy or has received treatment for a malignancy within the 12 months before Screening
14. Is currently receiving antipsychotic and/or selective serotonin reuptake inhibitor (SSRI) medications
15. Is receiving any other medication or has a condition that would preclude safe participation in the study or confound the evaluation of safety, as determined by the Investigator
16. Has a history of suicidal behavior (i.e., actions intended to harm oneself), suicidal ideation (ie, thoughts and plans about suicide), or suicide attempts
17. Has affirmative responses on the Columbia Suicide Severity Rating Scale (C-SSRS) questionnaire
18. Is currently taking supraphysiologic doses of systemic glucocorticoids for more than 3 weeks, except for intermittent short courses of exogenous glucocorticoids as needed for the treatment of asthma
19. Has received any other investigational compound within 1 month prior to screening or 5 half-lives of the investigational product (whichever is longer)
20. Has received gonadotropin-releasing hormone (GnRH) agonists, aromatase inhibitors, androgens (eg, dehydroepiandrosterone [DHEA]), anabolic steroids such as oxandrolone, or other sex steroids within 12 months before the Screening visit, or would require these treatments at any time during the study.
21. Receiving cytochrome P450 (CYP) 3A4 or P glycoprotein (P-gp) inhibitors/inducers or medications that are metabolized by CYP3A4 or P-gp within 30 days of enrolment.
22. Has a history of alcohol or drug abuse
23. Has a history or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, or other conditions that would preclude participation in the study, as determined by the Investigator
24. Has chronic urticaria or dermatographism
25. Has 25-hydroxy-vitamin D blood level < 20 ng/mL. Participants with initial vitamin D blood measurement < 20 ng/mL may receive supplementation per clinical practice during Screening and be rescreened up to 2 times

Ages: 12 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Increase in testosterone, as evaluated using PK parameters | From Enrollment through End of Study Assessments at Week 53

SECONDARY OUTCOMES:
Percentage of participants demonstrating either progression through Tanner Stages of puberty or attainment of Tanner Stage 5 by the end of the study | End of Study Assessment at Week 53
  Evaluated through clinical//physical examination
• Percentage of patients that had an increase in stretched penile length | End of Study Assessment at Week 53
  Evaluated through clinical//physical examination
Change from Screening or Baseline in DEXA bone density for total body less head (TBLH) and PA spine | End of Study Assessment at Week 53
  Evaluated through DEXA scan using age-appropriate software
Change from Screening or Baseline in body composition by DEXA scan | End of Study Assessment at Week 53
  Evaluated through DEXA scan using age-appropriate software
Change from Screening or Baseline in bone age as determined by X-ray | End of Study Assessment at Week 53
  Evaluated through X-ray using central readers
Change from Screening or Baseline in BMI-for-age percentile | End of Study Assessment at Week 53
  Evaluated through clinical//physical examination
• Change from Screening or Baseline in Height Velocity (HV) | End of Study Assessment at Week 53
  Evaluated through clinical//physical examination

OTHER OUTCOMES:
PK endpoints | End of Study Assessment at Week 53
  Total Testosterone concentration
Evaluation of Safety Endpoints including Treatment-Emergent Adverse Events | End of Study Assessment at Week 53
  Frequency and Severity of TEAEs

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Specialty Care - Jacksonville, Jacksonville, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - M Health Fairview U Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - The DOCS, Las Vegas, Nevada
  - Children's Hospital at Montefiore, The Bronx, New York
  - OUHSC Pediatric Diabetes & Endocrinology, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Prisma Health Children's Hospital - Midlands, Columbia, South Carolina
  - MedResearch, El Paso, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - MultiCare Institute for Research & Innovation, Tacoma, Washington